CLINICAL TRIAL: NCT05199662
Title: A Phase III, Randomized, Multi-center Clinical Trial That Will Examine Whether Treatment With Intravenous TNK is Superior to Placebo in Patients Who Suffer a Non-large Vessel Occlusion Ischemic Stroke Within 4.5-12 Hours From Time Last Seen Well
Brief Title: Randomization to Extend Stroke Intravenous ThromboLysis In Evolving Non-Large Vessel Occlusion With TNK (RESILIENT
Acronym: EXTEND-IV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Boehringer Ingelheim (Industry); Brainomix Limited (Industry); iSchemaView, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RESILIENT EXTEND-IV
Record Dates: First submitted 2021-12-13; First posted 2022-01-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke, Acute
Keywords: Ischemic Stroke; Thrombolysis; Tenecteplase
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Placebo administered as a single bolus injection over 5 seconds
  Interventions: Drug: Placebo
- Intravenous tenecteplase (TNK) (Experimental): Intravenous thrombolysis with Tenecteplase (TNK) at a dose of 0.25 mg/Kg (maximum 25mg, administered as a bolus over 5 seconds)
  Interventions: Drug: Intravenous tenecteplase

INTERVENTIONS:
Drug: Intravenous tenecteplase — Intravenous tenecteplase (TNK). Patients will receive intravenous TNK (0.25mg/kg, maximum 25mg, administered as a bolus over 5 seconds).
  Other Names: TNK; Metalyse
  Arms: Intravenous tenecteplase (TNK)
Drug: Placebo — Placebo matching IV TNK
  Arms: Control group

SUMMARY:
A phase III, randomized, multi-center clinical trial that will examine whether treatment with intravenous TNK is superior to placebo in patients who suffer a non-large vessel occlusion ischemic stroke within 4.5-12 hours from time last seen well. The randomization employs a 1:1 ratio of intravenous thrombolysis with Tenecteplase (TNK) versus placebo in patients who suffer a non-large vessel occlusion ischemic stroke between 4.5 and 12 hours from time last seen well (TLSW) and with a clinical-radiological mismatch or evidence of salvageable brain tissue on perfusion imaging.

DETAILED DESCRIPTION:
Prospective, multi-center, randomized, controlled, double blinded trial. The randomization employs a 1:1 ratio of intravenous thrombolysis with Tenecteplase (TNK) versus placebo in patients who suffer a non-large vessel occlusion ischemic stroke between 4.5 and 12 hours from time last seen well (TLSW) and with a clinical-radiological mismatch or evidence of salvageable brain tissue on perfusion imaging. Randomization will be done under a minimization process using age (≤70 vs. >70 years), baseline NIHSS (≤10 vs. >10), therapeutic window (4.5-9 or 9-12 hours after TLKW), randomization scenario and clinical site. For the primary endpoint, subjects will be followed for 90 days post-randomization.

The total sample size is 466 participants (233 in each arm). Interim analysis is planned with 40% and 67% of the total sample, with the possibility of stopping due to efficacy or futility, in addition to an adaptive design based on the conditional probability of a positive result.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke where patient is ineligible for IV thrombolytic treatment with Alteplase due to onset >4.5 hours and is ineligible for endovascular treatment under standard of care due to absence of proximal arterial occlusion (e.g. intracranial ICA, MCA-M1 and dominant M2 segments, and vertebrobasilar arteries).

   * Dominant M2 segment is defined is a division supplying >50% of the MCA territory vs co-dominant supplying 50% of the MCA territory vs non-dominant supplying <50% of the MCA territory.
2. No significant pre-stroke functional disability (mRS ≤2).
3. Age ≥18 years (no upper age limit).
4. Clinical or imaging mismatch evidence in distal artery territories, defined as one of the following scenarios (A, B or C):

   * Scenario A - all of the following:

     * Significant cortical neurological deficit (moderate to severe afasia, moderate to severe heminegligence, severe hemianopsia) with the addition or not of motor symptoms OR any motor deficit accompanied of cortical symptoms of any severity;
     * Contrast-enhanced CT of the head or head MRI with <50% involvement of the vascular territory corresponding to the clinical manifestation;
     * Arterial head angiotomography or arterial head angioMRI WITHOUT proximal intracranial artery occlusion that would require endovascular therapy (for example, ICA intracranial, MCA-M1 and M2 dominant segments and vertebral and basilar arteries)
   * Scenario B - all of the following:

     * NIHSS score ≥ 4 due to any neurologic deficits;
     * Non-contrast CT of the head or head MRI com <50% involvement of the vascular territory corresponding to the clinical manifestation;
     * Arterial head angioCT or arterial head MRI WITHOUT proximal intracranial artery occlusion that would require endovascular therapy (for example, ICA intracranial, MCA-M1 and M2 dominant segments and vertebral and basilar arteries)
     * Arterial head angioCT with distal occlusion on MIP or wedge-shaped lesion on parenchymography on the source-image of angiotomography OR CT perfusion with wedge-shaped cortical lesion.
   * Scenario C - all of the following:

     * NIHSS score ≥ 4 due to any neurologic deficits;
     * The presence of a Target Mismatch defined as:

       * Ischemic Core <50cc (defined on NCCT/CTP* or DWI MRI) *Volume NCCT can be used to exclude patients if the investigator believes that its volume assessment is more reliable that the CTP in any particular case.
       * Mismatch Volume (Tmax >6sec lesion - Core volume lesion) >10cc
       * Mismatch Ratio >1.4
5. Patient treatable within 4.5-12 hours of symptom onset. Symptoms onset is defined as point in time the patient was last seen well (at baseline). Treatment start is defined as initiation of IV TNK or placebo infusion.

   * Patients who have woken up with the symptoms and don't have a mismatch FLAIR-DWI according to the WAKE-UP Trial image criteria will have their window considered to be >4.5 hours. In this case, the time last seen well must have been 12 hours at most.
6. Informed consent obtained from patient or acceptable patient surrogate.

Exclusion Criteria:

1. Intracranial hemorrhage (ICH) identified by CT or MRI.
2. Rapidly improving symptoms, particularly if in the judgment of the managing clinician that the improvement is likely to result in the patient without eligibility criteria.
3. Pre-stroke mRS score of ≥ 2 (indicating previous disability)
4. Contra indication to imaging with MR or CT with contrast agents.
5. Infarct core >1/3 MCA territory qualitatively or >50 mL quantitatively (determined by DWI lesion on MR).
6. Participation in any investigational study in the previous 30 days
7. Any terminal illness such that patient would not be expected to survive more than 1 year).
8. Baseline platelet count < 100.000/µL
9. Woman of childbearing potential who is known to be pregnant or who has a positive pregnancy test on admission.
10. Previous stroke within last three months.
11. Recent past history or clinical presentation of ICH, subarachnoid hemorrhage (SAH), arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm other than meningioma.
12. Current use of oral anticoagulants and a prolonged prothrombin time (INR > 1.6).
13. Use of heparin, except for low dose subcutaneous heparin, in the previous 48 hours and a prolonged partial thromboplastin time exceeding the upper limit of the local laboratory normal range
14. Use of glycoprotein IIb - IIIa inhibitors within the past 72 hours. Use of single agent oral platelet inhibitors (clopidogrel or low-dose aspirin) prior to study entry is permitted.
15. Clinically significant hypoglycemia.
16. Uncontrolled hypertension defined by a blood pressure > 185 mmHg systolic or >110 mmHg diastolic on at least 2 separate occasions at least 10 minutes apart, or requiring aggressive treatment to reduce the blood pressure to within these limits. The definition of "aggressive treatment" is left to the discretion of the responsible Investigator.
17. Hereditary or acquired hemorrhagic diathesis.
18. Gastrointestinal or urinary bleeding within the preceding 21 days.
19. Major surgery within the preceding 14 days which poses risk in the opinion of the Investigator.
20. Exposure to a thrombolytic agent within the previous 72 hours.
21. Subject participating in a study involving an investigational drug or device that would impact this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rates of Good Functional Outcomes adjusted for the baseline mRS and stroke severity (NIHSS) according to the modified Rankin Scale scores at 90 days | 90 days
  Rates of Good Functional Outcomes adjusted for the baseline mRS and stroke severity (NIHSS) according to the modified Rankin Scale scores at 90 days as following:
  Baseline mRS=0 and NIHSS <10: mRs 90 days ≤1 Baseline mRS=1 and NIHSS ≥10: mRs 90 days ≤2

SECONDARY OUTCOMES:
Rates of Excellent Outcome defined as mRS ≤ 1 and/ or equal to Baseline mRS at 90 days | 90 days
  Rates of Excellent Outcome defined as mRS ≤ 1 and/ or equal to Baseline mRS at 90 days
Rates of Independent Outcome defined as mRS ≤ 2 and/ or equal to Baseline mRS at 90 days | 90 days
  Rates of Independent Outcome defined as mRS ≤ 2 and/ or equal to Baseline mRS at 90 days
Mean score for disability on the utility-weighted modified Rankin scale (UW-mRS) at 90 days | 90 days
  Mean score for disability on the utility-weighted modified Rankin scale (UW-mRS) at 90 days
Final infarct volume (FIV) and infarct growth (FIV - baseline infarct on CTP or DWI) evaluated on CT or MRI at 3-5 days (if available) | 3-5 days
  Final infarct volume (FIV) and infarct growth (FIV - baseline infarct on CTP or DWI) evaluated on CT or MRI at 3-5 days (if available)
Final infarct volume (FIV) and infarct growth (FIV - baseline infarct on CTP or DWI) evaluated on CT or MRI at 24 hours (-2/+12 hours) | 24 hours (-2/+12 hours)
  Final infarct volume (FIV) and infarct growth (FIV - baseline infarct on CTP or DWI) evaluated on CT or MRI at 24 hours (-2/+12 hours)
Dramatic early favorable response as determined by an NIHSS of 0-2 or NIHSS improvement ≥ 4 points at 24 (-2/+12 hours) hours | 24 (-2/+12 hours) hours
  Dramatic early favorable response as determined by an NIHSS of 0-2 or NIHSS improvement ≥ 4 points at 24 (-2/+12 hours) hours
Quality of life analysis as measured by EuroQol/EQ5D at 3 month, 6 months and one year, between interventional therapy vs medical therapy alone | 3 month, 6 months and one year
  Quality of life analysis as measured by EuroQol/EQ5D at 3 month, 6 months and one year, between interventional therapy vs medical therapy alone
Brain tissue reperfusion evaluated by CT or MRI perfusion at 24 hours in both treatment groups (if available) | 24 hours
  Brain tissue reperfusion evaluated by CT or MRI perfusion at 24 hours in both treatment groups (if available)
Mortality at 90 days ( safety outcome) | 90 days
  Mortality at 90 days ( safety outcome)
Clinically significant ICH rates at 24 (-2/+12) hours. | 24 (-2/+12) hours
  Clinically significant ICH rates at 24 (-2/+12) hours. All intracerebral hemorrhages will be classified by a central core-lab using the ECASS criteria. Symptomatic ICH will be defined as per the modified SITS-MOST definition: local or remote parenchymal hemorrhage type 2, subarachnoid hemorrhage, and/or intraventricular hemorrhage on the post-treatment imaging scan, combined with a neurological deterioration of 4 points or more on the NIHSS from baseline, or from the lowest NIHSS value between baseline and 24 h, or leading to death that the CEC/DSMB judges is causative of the deterioration.
Incidence of any intracranial hemorrhage (Heidelberg criteria) measured at 24 (-2/+12) | 24 (-2/+12)
  Incidence of any intracranial hemorrhage (Heidelberg criteria) measured at 24 (-2/+12) hours
Distribution of the modified Rankin Scale scores at 90 days (shift analysis) as evaluated by two separate assessors at the central core lab) who are blinded to treatment. | 90 days
  Distribution of the modified Rankin Scale scores at 90 days (shift analysis) as evaluated by two separate assessors at the central core lab) who are blinded to treatment. Primary Endpoint will consider central core lab readings only (video interview with RFA method) with local reading as a back-up mechanism

OTHER OUTCOMES:
Cost effectiveness analysis of IV TNK vs standard medical therapy | 12 months
  Cost effectiveness analysis of IV TNK vs standard medical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gisele Sampaio Silva, MD, MPH, PhD, Principal Investigator — Universidade Federal de São Paulo; Raul G Nogueira, MD, Principal Investigator — Emory University; Sheila CO Martins, MD, PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (14):
- Brazil (14):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas Botucatu, Botucatu
  - Hospital das Clínicas - UNICAMP, Campinas
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande
  - Hospital das Clínicas UFPR, Curitiba
  - Hospital Geral de Fortaleza, Fortaleza
  - Clinica Neurologica e Neurocirurgica de Joinville, Joinville
  - Hospital Metropolitano de Maceió, Maceió
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - Universidade de São Paulo, Ribeirão Preto
  - Hospital de Base São José do Rio Preto, São José do Rio Preto
  - Hospital São Paulo, São Paulo
  - Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Hospital Estadual Central, Vitória

IPD SHARING:
Plan to Share IPD: Undecided